CLINICAL TRIAL: NCT04322474
Title: Russian National Registry of Left Atrial Appendage Occlusion
Brief Title: Russian National Registry of LAAO
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 8-5
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; left atrial appendage; stroke prevention; occluder; Watchman device; Amplatzer Cardiac Plug
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Catheter-based left atrial appendage occlusion — Catheter-based implantation of left atrial appendage occluder

SUMMARY:
The first Russian registry presents data from two hundred consecutive patients with nonvalvular atrial fibrillation, who undergone left atrial appendage occlusion (LAAO) using the Watchman device and the Amplatzer cardiac plug. This government-funded catheter-based LAAO program was started in September 2015 and was completed in December 2017. Data collection was finished in December 2018. Five clinics agreed to participate in the study.

Patients' baseline characteristics, procedure, and follow up data were collected according to established registry protocol. Patients were followed at 45 days, 3, 6 and 12 months after enrollment. At each follow-up visit, the data regarding clinical events and healthcare utilization was collected.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years nonvalvular atrial fibrillation,
* CHA2DS2VASc ≥2,
* high risk of hemorrhagic events,
* non-compliance with pharmacological anticoagulant therapy

Exclusion Criteria:

* significant mitral valve disease,
* left ventricular ejection fraction <35%,
* the tendency to systemic thrombosis,
* severe co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonvalvular atrial fibrillation patients with a high risk of thromboembolic and haemorrhagic events
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Procedure-related major adverse events (pericardial effusion, cardiac tamponade, device embolization, procedure/device-related death) | 12 months
The composite of thromboembolic events, device thrombosis, hemorrhagic events, unexplained death | 12 months
  Primary efficacy endpoint

SECONDARY OUTCOMES:
Procedure success rate | intraprocedural
  successful left atrial appendage occluder implantation rate
Peridevice leakage | 6 months
  incidence rates of significant (≥5mm) leakage

CONTACTS AND LOCATIONS:
Overall Officials: Karapet Davtyan, PhD, Principal Investigator — National Research Center for Preventive Medicine